CLINICAL TRIAL: NCT03016767
Title: Efficacy of a Manual Oral Stimulation Protocol in Preterm Infants to Shorten the Period Between Enteral and Oral Nutrition
Brief Title: Efficacy of an Oral Stimulation Protocol in Preterm Infants to Shorten the Period Between Enteral and Oral Nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Para La Investigacion Hospital La Fe (Other)
Responsible Party: Principal Investigator, Marta Aguilar-Rodriguez, Dr., Fundacion Para La Investigacion Hospital La Fe
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014_0679_PP
Record Dates: First submitted 2016-12-30; First posted 2017-01-11 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Infant, Premature, Diseases
Keywords: oral feeding; oral stimulation; physiotherapy intervention
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- oral stimulation (Experimental): All the subjects of the study will receive the usual medical and nursing care for premature babies. They also will receive the physiotherapeutic treatment prescribed by the rehabilitation physician, focused mainly on respiratory and musculoskeletal care.
  Infants of the experimental group, in addition, will be applied a manual oral stimulation protocol designed ad hoc for this study, which consists of 12 maneuvers performed by a physiotherapist.
  Interventions: Procedure: Manual oral stimulation protocol
- non oral stimulation (No Intervention): All the subjects of the study will receive the usual medical and nursing care for premature babies. They also will receive the physiotherapeutic treatment prescribed by the rehabilitation physician, focused mainly on respiratory and musculoskeletal care. But this group will not be applied the oral stimulation protocol.

INTERVENTIONS:
Procedure: Manual oral stimulation protocol
  Arms: oral stimulation

SUMMARY:
Oral feeding in the neonatal period requires an accurate coordination between suction, swallowing and breathing. In premature new-borns and, depending on their gestational age, the coordinated work of those processes becomes jeopardised, being necessary to begin with an artificial enteral feeding. This situation results in lengthen their stay at the hospital until they are able to respond in a reliable way to their nutritional requirements orally, maintaining an adequate daily weight gain and without endangering their cardiorespiratory system.

This project is an experimental, prospective, blinded, randomized study, aimed to determine whether the application of a manual oral stimulation protocol in premature infants, hospitalized in a neonatal unit, reduces the transition time from enteral feeding to oral full feeding, while improves quality of feeding and shortens hospitalization time.

ELIGIBILITY:
Inclusion Criteria:

* Babies between 25 + 0 to 30 + 6 weeks of gestation according to the last menstruation, with adequate weight and size for their gestational age, who are receiving orogastric tube feeding, presenting clinical hemodynamic and cardiorespiratory stability and without any associated pathology.

Exclusion Criteria:

* Babies with congenital anomalies that affect feeding (chromosomopathies, craniofacial anomalies, severe esophageal or tracheal atresia, or any other that affect feeding),
* Babies with abnormalities that alter digestive function such as "necrotizing enterocolitis".
* Babies with other abnormalities that alter hemodynamic or cardiorespiratory stability, that present severe sepsis or positive meningitis culture, that suffer from chronic medical complications such as severe bronchopulmonary dysplasia, grade III or IV intraparaventricular hemorrhage, periventricular leukomalacia, etc.,
* Inability to to assign an exact gestational age.

Ages: 25 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
T1: Time elapsed, in days, from the end of the oral stimulation protocol (OSP) until the baby is able to ingest, through nutritive suction,100% of the total of the corresponding intake for his/her weight. | An average of 20 days after the baby is 32 weeks (32+0 to 32+6)
  A neonatology nurse, blinded to the study, routinely records, after each intake and on the habitual nursing evolution sheet, the amounts of milk that prematures take and the way of feeding (enteral, oral), among other factors (height, weight, percentile, incidences...). When the premature reaches 30 weeks of gestational age (30 + 0 to 30 + 6), the physiotherapist perform the ten-day manual oral stimulation protocol. The researchers will look at the nursing evolution sheet, the time (days) elapsed from the end of the protocol (equivalent day in control group) to the day in which babies are able to take 100% of the corresponding intake for their weight. Is estimated that experimental group will reach this goal approximately 3 days before than control group.
T2: Time elapsed, in days, from the end of the OSP until the baby is able to ingest, through nutritive suction, 30% of the total of the corresponding intake for his/her weight. | An average of 10 days after the baby is 32 weeks (32+0 to 32+6)
  30% suction without complications means that the baby already has the reflexes integrated and is able to coordinate suction, swallowing and breathing.
  A neonatology nurse, blinded to the study, routinely records, after each intake and on the habitual nursing evolution sheet, the amounts of milk that prematures take and the way of feeding (enteral, oral), among other factors (height, weight, percentile, incidences...). When the premature reaches 30 weeks of gestational age (30 + 0 to 30 + 6), the physiotherapist perform the ten-day manual oral stimulation protocol. The researchers will look at the nursing evolution sheet, the time (days) elapsed from the end of the protocol (equivalent day in control group) to the day in which babies are able to take 30% of the corresponding intake for their weight. Is estimated that experimental group will reach this goal approximately 4-5 days before than control group
T3: Time elapsed, in days, from the end of the OSP protocol until the baby is able to perform a full oral feeding, defined as the intake, by nutritive suction, of a quantity of milk ≥ 150 ml / kg / day , for three consecutive days. | An average of 25 days after the baby is 32 weeks (32+0 to 32+6)
  To be able to intake, by nutritive suction, of a quantity of milk ≥ 150 ml / kg / day , for three consecutive days (full oral feeding), is a discharge criterion in the Hospital la Fe of Valencia.
  A neonatology nurse, blinded to the study, routinely records, after each intake and on the habitual nursing evolution sheet, the amounts of milk that prematures take and the way of feeding (enteral, oral), among other factors (height, weight, percentile, incidences...). When the premature reaches 30 weeks of gestational age (30 + 0 to 30 + 6), the physiotherapist perform the ten-day manual oral stimulation protocol. The researchers will look at the nursing evolution sheet, the time (days) elapsed from the end of the protocol (equivalent day in control group) to the day in which babies are able to take a quantity of milk ≥ 150 ml / kg / day , for three consecutive days. Is estimated that experimental group will reach this goal approximately 4 days before than control group.
T4: Time of hospitalization of the babies. | An average of 9 weeks after the baby was hospitalized
  When babies are discharged from the hospital, researchers calculate the difference between gestational age (GE) the day they are discharged and the GE they were hospitalized. Is estimated that experimental group will reach this goal approximately 3 days before than control group.

SECONDARY OUTCOMES:
Weight gain of babies | When babies are discharged from the hospital, an average of 9 weeks after the babies were hospitalized
  Improving the weight gain of experimental group is also one of the main results in similar studies.
  When babies are discharged from the hospital, researchers look at the nursing evolution sheet, their weight gain (percentile) along their hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario y Politécnico La Fe, Valencia, Spain